CLINICAL TRIAL: NCT00358111
Title: A Single Arm Multi-Center Post Approval Study of LUMA as Adjunct to Colposcopy
Brief Title: Study of LUMA Cervical Imaging System as Adjunct to Colposcopy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PMA withdrawn
Sponsor: SpectraScience (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 302925
Record Dates: First submitted 2006-07-27; First posted 2006-07-28 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Dysplasia; Cancer
Keywords: high-grade disease; Cervical examination; targeting biopsies; dysplasia; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Luma Cervical Imaging System — Colposcopy using LUMA Cervical Imaging System

SUMMARY:
This is a post-approval, multi-center, single-arm study (n=950) designed to address the relationship of the LUMA device performance to patient age, patient human papillomavirus (HPV) status and colposcopist experience.

ELIGIBILITY:
Inclusion Criteria:

* Documented abnormal pap test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Relationship between HPV and the performance of the LUMA system as an adjunct to colposcopy for detection of CIN 2,3+ will be assessed. | ongoing - estimated at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jim Hitchin, Study Chair — SpectraScience
Locations (2):
- United States (2):
  - Women's Interventional Health, Encinitas, California
  - U of Iowa Health Center, Iowa City, Iowa